CLINICAL TRIAL: NCT04913207
Title: Comparison of Comprehensive CT-guided Versus Traditonal Echo-fluoroscopy-guided Strategy in the Implantation of the LAmbre Left Atrial Appendage Occlusion, a Prospective, Multi-center and Randomized Trial
Brief Title: Comprehensive CT-guided vs Echo-fluoroscopy-guided Strategy in the Left Atrial Appendage Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAAO-3DCT
Record Dates: First submitted 2021-05-27; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-03

CONDITIONS: Cardiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional echo-fluoroscopy guided group (Sham Comparator): LAA angiography is performed with a 6F pigtail catheter in LAA at the view of RAO 30°, CAU 20° and RAO 30°, CRA 20°. Next, the outline of the LAA will be drawn on the screen according to the LAA angiography. LAmbre device size selection is based on diameters of LAA ostium and landing zone measured on LAA angiography. The process of device implantation, assessment, releasing will be carried out at RAO 30°, CAU 20°. TEE is used to check whether the residual peri-device leaks is less than 5mm. The device will be released if it passes the 'COST' standard; otherwise readjusting the implantation position, change the device size and even re-puncturing transseptal to achieve a better axis will be proceeded.
  Interventions: Procedure: method of device size selection
- 3D-CTA guided group (Experimental): Patients in 3D-CTA based perimeter group will undergo CCTA examination before LAAO and a 3D model of the left atrium is reconstructed by a workstation. LAmbre device size selection is based on perimeters of LAA ostium and landing zone which are obtained by the measurement method shown previously in this protocol. After transseptal puncture, LAA angiography is performed with a 6F pigtail catheter in LAA at the tangent angle view which is obtained preoperatively by 3D-CCTA. Then, the outline of the LAA will be drawn on the screen according to the LAA angiography. The process of device implantation, assessment, releasing will be carried out at this tangent angle view. TEE is used to check whether the residual peri-device leaks is less than 5mm. The device will be released if it passes the 'COST' standard; otherwise readjusting the implantation position, change the device size and even re-puncturing transseptal to achieve a better axis will be proceeded.
  Interventions: Procedure: method of device size selection

INTERVENTIONS:
Procedure: method of device size selection — device size selection based on 3D-CTA

SUMMARY:
Percutaneous left atrial appendage occlusion (LAAO) is an increasingly used alternative to oral anticoagulation in patients with nonvalvular atrial fibrillation (AF). Transesophageal echocardiography (TEE) and fluoroscopy were used to measure the maximal diameters of LAA. However, the LAA maximal diameters measured on Two dimensional (2D) views could be limited due to the morphology of LAA varies with each individua. Three dimension computed tomography angiography technology (3D-CTA) is based on cardiac computed tomography angiography (CCTA). The 3D-CTA technology provides an innovative measuring method of LAA to guide the selection of device size, and the best fluoroscopy view to implant device. This measuring method and guideline have never been reported and its role in LAAO is uncertain

DETAILED DESCRIPTION:
The PERIVISION-LAAO study will be a prospective, multi-center and randomized trial designed to investigate the effect and safety of perimeter obtained by 3D-CTA versus diameter obtained by traditional echo-fluoroscopy in guidance of device size selection in the procedure of LAAO. It will enroll 310 patients with nonvalvular atrial fibrillation (AF) who will be randomized at 1:1 ratio into the perimeter guidance group or diameter guidance group. The major effect endpoint will be the success at first device selected in procedure, and the major safety outcome will be the incidence of pericardial effusion during the procedure and the follow-up period of 2 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of atrial fibrillation Disease
* Age >18years
* CHA2DS2-VASc scores ≥ 2
* And at least one of the following indications: (a) HAS- BLED scores ≥ 3; (b) intolerance to long-term OAC; (c) stroke, TIA or thromboembolism even under OAC treatment

Exclusion Criteria:

* GFR <50 mL/min/1.73 m2
* Thrombus in LA and LAA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of success at first device selected | In the procedure of LAAO
  the device selected successfully at first time during LAAO

CONTACTS AND LOCATIONS:
Overall Officials: HJ LUO, Study Chair — Shanghai Jiao Tong University, School of Medicine, Affiliated Ren Ji Hospital
Locations (1):
- Shanghai Jiao Tong University, School of Medicine, Affiliated Ren Ji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No